CLINICAL TRIAL: NCT00109551
Title: Zinc Supplementation Impact on Child Mortality--Nepal
Brief Title: Community Trial of Zinc Supplementation on Preschool Child Mortality and Morbidity in Southern Nepal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: R01HD038753 (NIH); R01HD038753 (NIH)
Record Dates: First submitted 2005-04-28; First posted 2005-04-29 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2006-01

CONDITIONS: Nutrition
Keywords: zinc; child mortality; child morbidity; community trial; prevention trial; dietary supplement

INTERVENTIONS:
Drug: zinc sulphate dietary supplement
Drug: iron sulphate-folic acid dietary supplement

SUMMARY:
The purpose of this study is to determine whether daily supplementation of young children in Nepal with either zinc, iron-folic acid, or both can reduce mortality and morbidity. Young children in Nepal have numerous nutritional deficiencies and high rates of morbidity and mortality. Zinc and/or iron supplementation may be a cost-effective method for reducing these risks.

DETAILED DESCRIPTION:
Mortality rates among preschool age children in Nepal and many other developing countries remain high despite significant progress made over the past 20 years. There remain significant nutritional deficiencies in these populations, especially important are vitamin and mineral deficiencies.

Comparisons: In this study, we are comparing the morbidity and mortality experience for children 1-36 months of age randomized to one of four daily supplementation regimens: placebo, zinc alone, iron-folic acid alone, zinc + iron-folic acid.

ELIGIBILITY:
Inclusion Criteria:

* All children 1-35 months of age living in 30 Village Development Committees of Sarlahi District in southern Nepal.

Exclusion Criteria:

* Parent refusal

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58000
Dates: Start 2001-10; Study Completion 2006-01

PRIMARY OUTCOMES:
Death among children 1-36 months of age

SECONDARY OUTCOMES:
Incidence rates of selected morbidities including diarrhea, dysentery, acute respiratory infections

CONTACTS AND LOCATIONS:
Overall Officials: James M Tielsch, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (3):
- United States (2):
  - Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - Cornell University Division of Nutritional Sciences, Ithaca, New York
- Nepal Nutrition Intervention Project-Sarlahi, Kathmandu and Sarlahi District, Nepal

REFERENCES:
- [Result] Tielsch JM, Khatry SK, Stoltzfus RJ, Katz J, LeClerq SC, Adhikari R, Mullany LC, Shresta S, Black RE. Effect of routine prophylactic supplementation with iron and folic acid on preschool child mortality in southern Nepal: community-based, cluster-randomised, placebo-controlled trial. Lancet. 2006 Jan 14;367(9505):144-52. doi: 10.1016/S0140-6736(06)67963-4. PMID 16413878
- [Result] Coles CL, Sherchand JB, Khatry SK, Katz J, Leclerq SC, Mullany LC, Tielsch JM. Nasopharyngeal carriage of S. pneumoniae among young children in rural Nepal. Trop Med Int Health. 2009 Sep;14(9):1025-33. doi: 10.1111/j.1365-3156.2009.02331.x. Epub 2009 Jun 28. PMID 19563428
- [Result] Kordas K, Siegel EH, Olney DK, Katz J, Tielsch JM, Kariger PK, Khalfan SS, LeClerq SC, Khatry SK, Stoltzfus RJ. The effects of iron and/or zinc supplementation on maternal reports of sleep in infants from Nepal and Zanzibar. J Dev Behav Pediatr. 2009 Apr;30(2):131-9. doi: 10.1097/DBP.0b013e31819e6a48. PMID 19322104
- [Result] Coles CL, Sherchand JB, Khatry SK, Katz J, Leclerq SC, Mullany LC, Tielsch JM. Zinc modifies the association between nasopharyngeal Streptococcus pneumoniae carriage and risk of acute lower respiratory infection among young children in rural Nepal. J Nutr. 2008 Dec;138(12):2462-7. doi: 10.3945/jn.108.095422. PMID 19022973
- [Result] Kordas K, Siegel EH, Olney DK, Katz J, Tielsch JM, Chwaya HM, Kariger PK, Leclerq SC, Khatry SK, Stoltzfus RJ. Maternal reports of sleep in 6-18 month-old infants from Nepal and Zanzibar: association with iron deficiency anemia and stunting. Early Hum Dev. 2008 Jun;84(6):389-98. doi: 10.1016/j.earlhumdev.2007.10.007. Epub 2007 Nov 26. PMID 18022771
- [Result] Tielsch JM, Khatry SK, Stoltzfus RJ, Katz J, LeClerq SC, Adhikari R, Mullany LC, Black R, Shresta S. Effect of daily zinc supplementation on child mortality in southern Nepal: a community-based, cluster randomised, placebo-controlled trial. Lancet. 2007 Oct 6;370(9594):1230-9. doi: 10.1016/S0140-6736(07)61539-6. PMID 17920918
- [Result] Siegel EH, Stoltzfus RJ, Khatry SK, Leclerq SC, Katz J, Tielsch JM. Epidemiology of anemia among 4- to 17-month-old children living in south central Nepal. Eur J Clin Nutr. 2006 Feb;60(2):228-35. doi: 10.1038/sj.ejcn.1602306. PMID 16234835
- [Result] Siegel EH, Stoltzfus RJ, Kariger PK, Katz J, Khatry SK, LeClerq SC, Pollitt E, Tielsch JM. Growth indices, anemia, and diet independently predict motor milestone acquisition of infants in south central Nepal. J Nutr. 2005 Dec;135(12):2840-4. doi: 10.1093/jn/135.12.2840. PMID 16317129
- [Result] Katz J, Khatry SK, Leclerq SC, Mullany LC, Yanik EL, Stoltzfus RJ, Siegel EH, Tielsch JM. Daily supplementation with iron plus folic acid, zinc, and their combination is not associated with younger age at first walking unassisted in malnourished preschool children from a deficient population in rural Nepal. J Nutr. 2010 Jul;140(7):1317-21. doi: 10.3945/jn.109.119925. Epub 2010 May 19. PMID 20484548
- [Result] Wu L, Katz J, Mullany LC, Haytmanek E, Khatry SK, Darmstadt GL, West KP Jr, LeClerq SC, Tielsch JM. Association between nutritional status and positive childhood disability screening using the ten questions plus tool in Sarlahi, Nepal. J Health Popul Nutr. 2010 Dec;28(6):585-94. doi: 10.3329/jhpn.v28i6.6607. PMID 21261204
- [Result] Wu LA, Katz J, Mullany LC, Khatry SK, Darmstadt GL, LeClerq SC, Tielsch JM. The association of preterm birth and small birthweight for gestational age on childhood disability screening using the Ten Questions Plus tool in rural Sarlahi district, southern Nepal. Child Care Health Dev. 2012 May;38(3):332-40. doi: 10.1111/j.1365-2214.2011.01221.x. Epub 2011 Mar 6. PMID 21375569
- [Result] Siegel EH, Kordas K, Stoltzfus RJ, Katz J, Khatry SK, LeClerq SC, Tielsch JM. Inconsistent effects of iron-folic acid and/or zinc supplementation on the cognitive development of infants. J Health Popul Nutr. 2011 Dec;29(6):593-604. doi: 10.3329/jhpn.v29i6.9896. PMID 22283033
- [Result] Surkan PJ, Shankar M, Katz J, Siegel EH, Leclerq SC, Khatry SK, Stoltzfus RJ, Tielsch JM. Beneficial effects of zinc supplementation on head circumference of Nepalese infants and toddlers: a randomized controlled trial. Eur J Clin Nutr. 2012 Jul;66(7):836-42. doi: 10.1038/ejcn.2012.42. Epub 2012 May 9. PMID 22569086
- [Result] Surkan PJ, Siegel EH, Patel SA, Katz J, Khatry SK, Stoltzfus RJ, Leclerq SC, Tielsch JM. Effects of zinc and iron supplementation fail to improve motor and language milestone scores of infants and toddlers. Nutrition. 2013 Mar;29(3):542-8. doi: 10.1016/j.nut.2012.09.003. Epub 2013 Jan 5. PMID 23298972
- [Derived] Surkan PJ, Charles MK, Katz J, Siegel EH, Khatry SK, LeClerq SC, Stoltzfus RJ, Tielsch JM. The role of zinc and iron-folic acid supplementation on early child temperament and eating behaviors in rural Nepal: a randomized controlled trial. PLoS One. 2015 Mar 30;10(3):e0114266. doi: 10.1371/journal.pone.0114266. eCollection 2015. PMID 25821959
- [Derived] Christian P, Morgan ME, Murray-Kolb L, LeClerq SC, Khatry SK, Schaefer B, Cole PM, Katz J, Tielsch JM. Preschool iron-folic acid and zinc supplementation in children exposed to iron-folic acid in utero confers no added cognitive benefit in early school-age. J Nutr. 2011 Nov;141(11):2042-8. doi: 10.3945/jn.111.146480. Epub 2011 Sep 28. PMID 21956955